CLINICAL TRIAL: NCT01120249
Title: EVEREST: EVErolimus for Renal Cancer Ensuing Surgical Therapy, A Phase III Study
Brief Title: S0931, Everolimus in Treating Patients With Kidney Cancer Who Have Undergone Surgery
Acronym: S0931
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S0931; S0931 (Other: SWOG); U10CA032102 (NIH); NCI-2011-02028 (Other: NCI)
Record Dates: First submitted 2010-05-07; First posted 2010-05-10 (Estimated); Results first posted 2024-03-20 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; clear cell renal cell carcinoma; papillary renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral everolimus once daily on days 1-42. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus
- Arm II (Placebo Comparator): Patients receive oral placebo once daily on days 1-42. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: everolimus — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor.

PURPOSE: This phase III trial is studying everolimus to see how well it works in treating patients with kidney cancer who have undergone surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* to compare recurrence-free survival in renal carcinoma patients randomly assigned to 54 weeks of everolimus versus 54 weeks of placebo after nephrectomy or partial nephrectomy.

Secondary

* To compare the overall survival of patients treated with everolimus vs placebo.
* To compare qualitative and quantitative toxicity between the two study arms.
* To bank tissue and biologic specimens for future study of molecular biomarkers relevant to the AKT/mTOR and other pathways implicated in the pathogenesis of renal carcinoma and to investigate their potential predictive and prognostic value.
* To bank blood specimens for the future study of the relationship between steady-state trough levels of everolimus and relevant side effects (lymphopenia, infection, hyperglycemia, hypercholesterolemia, hypertriglyceridemia) in patients treated on this study with everolimus.

OUTLINE: This is a multicenter study.

Patients are stratified according to pathologic stage (intermediate high-risk vs very high-risk), histologic subtype (clear cell vs non-clear cell), and performance status (0 vs 1). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral everolimus once daily on days 1-42. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo once daily on days 1-42. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.

Archived tumor tissue, plasma, and whole blood samples may be collected periodically for biomarker analysis and other translational studies.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually for 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma

  * Clear cell or non-clear cell allowed

    * No disease of the collecting duct or medullary carcinoma
  * Considered pathologically either intermediate high-risk or very high-risk disease
  * No history of distant metastases
  * Patients with microvascular invasion of the renal vein of any grade or stage (as long as M0) are eligible
* Have undergone a full surgical resection (radical nephrectomy or partial nephrectomy) including removal of all clinically positive nodes

  * Surgical margins must be negative

    * Patients with positive renal vein margins are eligible unless there is invasion of the renal vein wall at the margin (provided no other margins are positive)
  * Patients must be registered within 84 days after the date of the first surgical resection of the first tumor
* No evidence of residual or metastatic renal cell cancer on CT scan of the chest, abdomen, and pelvis (all with oral and IV contrast) performed after nephrectomy and within 28 days before registration

  * MRI scans of the abdomen and pelvis with gadolinium and a non-contrast CT scan of the chest may be substituted if the patient is not able to have CT scans with IV contrast

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 2.0 times upper limit of normal (ULN) OR calculated creatinine clearance ≥ 30 mL/min
* Bilirubin ≤ 1.5 times ULN
* SGOT and SGPT ≤ 2.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for up to 8 weeks after completion of study treatment
* Able to take oral medications
* Patients must not have any of the following:

  * NYHA class III-IV cardiac disease (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort)
  * Unstable angina pectoris
  * Myocardial infarction within the past 6 months
  * Serious uncontrolled cardiac arrhythmia
* Patients must NOT have liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh Class C)
* HBV and HCV testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection
* Must be able to take oral medications
* No impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* No known history of HIV seropositivity
* No known uncontrolled, underlying pulmonary disease (spirometry and DLCO ≤ 50% of predicted OR oxygen saturation ≤ 88% at rest on room air)
* No uncontrolled hyperlipidemia (fasting serum cholesterol > 300 mg/dL AND fasting triglycerides > 2.5 times ULN) obtained within 28 days prior to registration

  * Optimal lipid control must be achieved before registration and monitored during protocol treatment
* No uncontrolled diabetes mellitus (defined by fasting serum glucose > 1.5 times ULN) obtained within 28 days prior to registration.

  * Optimal glucose control must be achieved before registration and monitored during protocol treatment
* No prior malignancies except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or stage II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years
* No known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to their excipients
* No contraindications to receiving either IV iodine-based contrast or gadolinium

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Patients must have recovered from any surgery-related complications
* No prior anticancer therapy for renal cell carcinoma including systemic therapy in the adjuvant or neoadjuvant setting, immunotherapy, investigational therapy, surgical metastasectomy, or radiotherapy
* More than 14 days since prior and no concurrent strong CYP3A4 inhibitors (i.e., ketoconazole, itraconazole, voriconazole, posaconazole, fluvoxamine, nefazodone, nelfinavir, or ritonavir) or strong CYP3A4 inducers (i.e., phenytoin, rifampin, or rifabutin)
* More than 7 days since prior and no concurrent live vaccines
* No other concurrent anticancer agents including investigational agents
* No concurrent chronic treatment with systemic steroids or another immunosuppressive agent

  * Topical or inhaled corticosteroids are allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1545 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W. Ryan, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1003):
- United States (1002):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Gulf Coast MBCCOP, Mobile, Alabama
  - Providence Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Cancer Center at UMC Orange Grove, Tucson, Arizona
  - Arizona Cancer Center at University Medical Center North, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veteran's Administration Medical Center, Little Rock, Arkansas
  - Kaiser Anaheim Medical Center, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente Medical Group - Baldwin Park, Baldwin Park, California
  - Kaiser Foundation Hospital, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Northbay Cancer Center, Fairfield, California
  - Kaiser Permanente Hospital, Fontana, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Saint Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Southern California Permanente Medical Group, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-West Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Epic Care-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente Medical Center, Riverside, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-Mission, San Diego, California
  - Kaiser Permanente at San Diego, San Diego, California
  - Kaiser Permanente, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente Health Care, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Atlo Medical Foundation-Sunnyvale, Sunnyvale, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Denver Veterans Administration Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - University of Connecticut, Farmington, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Florida Hospital Cancer Institute Altamonte, Altamonte Springs, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Florida Hospital Kissimmee, Kissimmee, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Florida Urology Associates-Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Florida Hospital East Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Sacred Heart Medical Oncology Group - Davis Highway, Pensacola, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Florida Hospital Cancer Institute Winter Park, Winter Park, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Leeward Radiation Oncology Center, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Resurrection Healthcare, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Central Illinois CCOP, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Galesburg Cottage Plaza Office, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Cadence Cancer Center at Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Adventist La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology-PC Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Promise Regional Medical Center-Hutchinson, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas City Cancer Center-West, Kansas City, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center-Shawnee Mission, Shawnee Mission, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Louisiana State University Sciences Center- Monroe, Monroe, Louisiana
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - York Hospital, York Village, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Veterans Administration Medical Center-Baltimore, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - The Memorial Hospital at Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Associates In Oncology Hematology PC-Rockville, Rockville, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Caritas Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren-Bay Region, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Great Lakes Cancer Institute, Clarkston, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Great Lakes Cancer Institute-Lapeer Campus, Lapeer, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Northern Michigan Regional Hospital, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Forest General Hospital, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Saint Francis Medical Center, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - Good Samaritan Hospital, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hemotology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Sunrise, Las Vegas, Nevada
  - Children's Specialty Center of Nevada II, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Alpine Hematology-Oncology, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Reno Oncology Consultants, Reno, Nevada
  - New Hampshire Oncology-Hematology PA, Concord, New Hampshire
  - New Hampshire Oncology Hematology Associates, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Cancer Institute of New Jersey At Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Kennedy Health Systems-Cancer Center, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Mountain Radiation Oncology, Asheville, North Carolina
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Transylvania Regional Hospital, Brevard, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Carolinas Medical Center - Northeast, Concord, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Lexington, North Carolina
  - McDowell Hospital, Marion, North Carolina
  - Carolinas Medical Center-Union, Monroe, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Cleveland Regional Medical Center, Shelby, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Southeast Cancer Control Consortium CCOP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology and Hematology Care Inc-Taft, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Summa Health Center at Lake Medina, Medina, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Mercy, Oklahoma City, Oklahoma
  - Oklahoma Oncology Inc, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Cancer Research Foundation, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Saint Charles Medical Center-Bend, Bend, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Health System, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - UPMC - HVHS Cancer Center at Heritage Valley Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - UPMC Cancer Center at Jefferson Regional Medical Center, Clairton, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Medical Oncology at Evangelical Community Hospital, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC-Uniontown/Robert E. Eberly Pavilion, Uniontown, Pennsylvania
  - Washington Hospital, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-Charleston, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Conklin Regional Cancer Center, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Kingsport, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Saint Luke's Episcopal Hospital, Houston, Texas
  - Veterans Administration Medical Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Danville Hematology Oncology, Danville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology Associates PC, Winchester, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Auburn Regional Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Aurora Cancer Care-Burlington, Burlington, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora Cancer Care-Southern Lakes, Elkhorn, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Advanced Healthcare Inc-Menomonee Falls, Menomonee Falls, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Wheaton Franciscan Healthcare - Saint Joseph, Milwaukee, Wisconsin
  - Aurora Cancer Care-Milwaukee South, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Waukesha Memorial Hospital - ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - The Alyce and Elmore Kraemer Cancer Care Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gulati S, Tangen C, Ryan CW, Vaishampayan UN, Shuch BM, Barata PC, Pruthi DK, Bergerot CD, Tripathi A, Lerner SP, Thompson IM Jr, Lara PN Jr, Pal SK. Adjuvant Everolimus in Non-Clear Cell Renal Cell Carcinoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2425288. doi: 10.1001/jamanetworkopen.2024.25288. PMID 39106067
- [Derived] Ryan CW, Tangen CM, Heath EI, Stein MN, Meng MV, Alva AS, Pal SK, Puzanov I, Clark JI, Choueiri TK, Agarwal N, Uzzo RG, Haas NB, Synold TW, Plets M, Vaishampayan UN, Shuch BM, Thompson IM Jr, Lara PN Jr. Adjuvant everolimus after surgery for renal cell carcinoma (EVEREST): a double-blind, placebo-controlled, randomised, phase 3 trial. Lancet. 2023 Sep 23;402(10407):1043-1051. doi: 10.1016/S0140-6736(23)00913-3. Epub 2023 Jul 28. PMID 37524096
- See also: Related Info — https://nctn-data-archive.nci.nih.gov/
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1545 total participants were randomly assigned; 770 on the placebo arm and 775 on the everolimus arm. 46 participants were deemed ineligible. Reasons for ineligibility include insufficient imaging or unable to rule out residual or metastatic disease, evidence of residual or metastatic disease, not intermediate-high or very-high risk, other active or recent cancer, and ineligible histology. This leaves 1499 eligible participants (744 placebo, 755 everolimus).
Groups:
- Placebo: Patients receive oral placebo once daily on days 1-42. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.
- Everolimus: Patients receive oral everolimus once daily on days 1-42. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Placebo | Everolimus
Started | 744 | 755
Completed | 512 | 343
Not Completed | 232 | 412
Not completed — No protocol treatment received | 21 | 15
Not completed — Disease recurrence | 107 | 57
Not completed — Death | 1 | 0
Not completed — Adverse Event | 40 | 276
Not completed — Participant refusal | 34 | 42
Not completed — Other reasons, not protocol specified | 29 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Everolimus | Total
Number analyzed (Participants) | 744 | 755 | 1499
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [50 to 66] | 58 [51 to 66] | 58 [51 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 235 | 457
  Male | 522 | 520 | 1042
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 670 | 688 | 1358
  Race: Black | 27 | 34 | 61
  Race: Asian | 20 | 11 | 31
  Race: Other/unknown | 27 | 22 | 49
Zubrod Performance Status [Count of Participants; unit: Participants] — A performance status of 0 is defined as fully active, able to carry on all pre-disease performance without restriction.
  A performance status of 1 is defined as restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Participants
    0 | 588 | 603 | 1191
    1 | 156 | 152 | 308
Risk Group [Count of Participants; unit: Participants]
  Intermediate-high | 337 | 343 | 680
  Very high | 407 | 412 | 819
Pathological T Stage [Count of Participants; unit: Participants] — pT1 - Tumor invades subepithelial connective tissue pT2 - Tumor invades muscularis pT3 - Tumor invades beyond muscularis into: peripelvic fat and renal parenchyma pT4 - Tumor invades adjacent organs OR through the kidney into perinephric fat pTX- Primary tumor cannot be assessed
  Participants
    pT1 | 71 | 62 | 133
    pT2 | 158 | 147 | 305
    pT3 | 498 | 525 | 1023
    pT4 | 14 | 17 | 31
    pTX | 3 | 4 | 7
Nephrectomy [Count of Participants; unit: Participants]
  Radical | 662 | 689 | 1351
  Partial | 82 | 66 | 148
Histology [Count of Participants; unit: Participants]
  Clear Cell | 622 | 626 | 1248
  Non-clear cell, Papillary | 52 | 57 | 109
  Non-clear cell, Chromophobe | 46 | 53 | 99
  Non-clear cell, Other | 24 | 19 | 43
Pathological Lymph Node Status [Count of Participants; unit: Participants] — pN0 - No regional lymph node metastasis pN+ (fully resected) - Metastasis in regional lymph node(s) pNx (clinically N0) - Regional lymph nodes cannot be assessed
  Participants
    pN0 | 220 | 219 | 439
    pN+ (fully resected) | 57 | 58 | 115
    pNx (clinically N0) | 467 | 478 | 945

OUTCOME MEASURES:

1. Primary Outcome: 5-year Recurrence-free Survival (RFS)
Description: To compare 5-year recurrence-free survival in renal carcinoma participants randomly assigned to 54 weeks of everolimus versus 54 weeks of placebo after nephrectomy or partial nephrectomy. Recurrence-free survival is defined as From date of registration to date of first documentation of recurrence or death due to any cause. Participants last known to be alive and recurrence-free are censored at date of last contact. Recurrence is defined as positive cytology or biopsy and/or progressively enlarging solid mass as evidenced by CT or MRI scans.
Time Frame: 5 years from registration
Population: 1545 total participants were randomly assigned; 770 on the placebo arm and 775 on the everolimus arm. 46 participants were deemed ineligible. Reasons for ineligibility include insufficient imaging or unable to rule out residual or metastatic disease, evidence of residual or metastatic disease, not intermediate-high or very-high risk, other active or recent cancer, and ineligible histology. This leaves 1499 eligible participants (744 placebo, 755 everolimus).
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | Placebo | Everolimus
Number analyzed (Participants) | 744 | 755
percentage of paticipants | 63 [60 to 67] | 67 [63 to 70]

2. Secondary Outcome: 5-year Overall Survival (OS)
Description: To compare 5-year overall survival in those patients randomized to everolimus versus those randomized to placebo. Overall survival is defined as time from date of registration to date of death due to any cause or patients last known to be alive are censored at their last contact date.
Time Frame: 5 years from registration
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | Placebo | Everolimus
Number analyzed (Participants) | 744 | 755
percentage of paticipants | 85 [82 to 87] | 87 [84 to 89]

3. Secondary Outcome: Frequency and Severity of Toxicities
Description: Number of participants with Grade 3-5 adverse events that are possibly, probably or definitely related to study drug are reported. Measured using CTCAE v4.0.
Time Frame: Up to 54 weeks of treatment
Population: Participants who received at least one dose of protocol treatment and were not excluded from safety analysis per the study chairs request.
Measure: Number; unit: Participants
Arm/Group | Placebo | Everolimus
Number analyzed (Participants) | 723 | 740
Participants
  Abdominal infection | 0 | 1
  Abdominal pain | 0 | 7
  Acidosis | 1 | 0
  Acute kidney injury | 2 | 2
  Agitation | 1 | 0
  Alanine aminotransferase increased | 3 | 6
  Allergic reaction | 0 | 1
  Anemia | 0 | 12
  Anorexia | 0 | 4
  Aortic valve disease | 0 | 1
  Arthralgia | 2 | 0
  Aspartate aminotransferase increased | 2 | 3
  Back pain | 1 | 2
  Bone infection | 0 | 2
  Bullous dermatitis | 0 | 1
  Cholesterol high | 2 | 2
  Chronic kidney disease | 1 | 3
  Colitis | 0 | 2
  Colonic perforation | 1 | 0
  Creatinine increased | 2 | 2
  Dehydration | 3 | 8
  Diarrhea | 5 | 11
  Dizziness | 1 | 0
  Dry skin | 0 | 5
  Dyspepsia | 1 | 0
  Dyspnea | 1 | 6
  Edema limbs | 0 | 3
  Endocarditis infective | 0 | 1
  Eye disorders - Other, specify | 1 | 0
  Fatigue | 5 | 27
  Gastritis | 1 | 0
  Gastrointestinal disorders - Other, specify | 1 | 1
  Generalized muscle weakness | 0 | 1
  Glucose intolerance | 0 | 2
  Headache | 1 | 2
  Heart failure | 0 | 2
  Hemorrhoids | 0 | 1
  Hoarseness | 1 | 0
  Hypercalcemia | 1 | 1
  Hyperglycemia | 3 | 37
  Hyperkalemia | 1 | 4
  Hypertension | 20 | 31
  Hypertriglyceridemia | 13 | 85
  Hyperuricemia | 1 | 1
  Hypokalemia | 1 | 0
  Hyponatremia | 1 | 4
  Hypophosphatemia | 1 | 2
  Hypotension | 0 | 1
  Hypoxia | 0 | 1
  INR increased | 0 | 1
  Immune system disorders - Other, specify | 0 | 1
  Infections and infestations - Other, specify | 1 | 3
  Irritability | 0 | 1
  Laryngeal mucositis | 0 | 1
  Leukocytosis | 0 | 1
  Localized edema | 0 | 1
  Lung infection | 1 | 5
  Lymphocyte count decreased | 1 | 5
  Mucositis oral | 2 | 103
  Multi-organ failure | 1 | 1
  Myocardial infarction | 0 | 1
  Nail infection | 0 | 1
  Nausea | 3 | 0
  Nervous system disorders - Other, specify | 0 | 1
  Neutrophil count decreased | 2 | 4
  Non-cardiac chest pain | 1 | 2
  Obesity | 1 | 1
  Pain | 0 | 2
  Pain in extremity | 0 | 2
  Peripheral sensory neuropathy | 1 | 0
  Photosensitivity | 2 | 0
  Pneumonitis | 0 | 9
  Proteinuria | 0 | 2
  Pruritus | 1 | 7
  Rash acneiform | 0 | 16
  Rash maculo-papular | 0 | 15
  Rash pustular | 0 | 1
  Renal and urinary disorders - Other, specify | 0 | 3
  Resp, thoracic and mediastinal disorders - Other | 0 | 3
  Seroma | 0 | 1
  Sinusitis | 0 | 1
  Skin and subcutaneous tissue disorders - Other | 1 | 0
  Skin infection | 1 | 3
  Soft tissue infection | 0 | 1
  Syncope | 2 | 2
  Thromboembolic event | 0 | 4
  Tooth infection | 0 | 2
  Upper respiratory infection | 0 | 1
  Urinary tract infection | 2 | 1
  Vomiting | 2 | 3
  Weight gain | 1 | 0
  Wheezing | 0 | 1
  Wound infection | 0 | 2

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 10 years post registration
Description: 1,463 eligible participants who received at least one dose of protocol treatment were evaluable for Adverse Events (AEs): 740 on the Everolimus arm and 723 on the placebo arm. AEs and Serious Adverse Events (SAEs) are reported by CTCAE Version 4.0.
Groups:
- Placebo: Patients receive oral placebo once daily on days 1-42. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity. Of the 770 participants assigned to this arm, 744 were eligible for efficacy analysis and included in the at-risk for all cause mortality population. The 723 participants who received placebo are included in at-risk for adverse event population.
- Everolimus: Patients receive oral everolimus once daily on days 1-42. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity. Of the 775 participants assigned to this arm, 755 were eligible for efficacy analysis and included in the at-risk for all cause mortality population. The 740 participants who received everolimus are included in at-risk for adverse event population.
Arm/Group | Placebo | Everolimus
All-Cause Mortality (participants affected / at risk) | 151/744 | 139/755
Serious Adverse Events (participants affected / at risk) | 68/723 | 154/740
Other Adverse Events (participants affected / at risk) | 649/723 | 716/740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=723) | Everolimus (N=740)
Anemia (Blood and lymphatic system disorders) | 3 | 8
Aortic valve disease (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac disorders-Other (Cardiac disorders) | 1 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 2
Heart failure (Cardiac disorders) | 1 | 3
Myocardial infarction (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 2
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Eye disorders-Other (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 10
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 2 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 8
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 22
Nausea (Gastrointestinal disorders) | 3 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5
Chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 3
Edema trunk (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 10
Fever (General disorders) | 1 | 3
General disorders and admin site conditions - Other (General disorders) | 0 | 2
Irritability (General disorders) | 0 | 1
Localized edema (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 6
Pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Immune system disorders-Other (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bone infection (Infections and infestations) | 0 | 2
Endocarditis infective (Infections and infestations) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 1 | 5
Lung infection (Infections and infestations) | 4 | 6
Nail infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 2
Tooth infection (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 4 | 0
Wound infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Cardiac troponin I increased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 4 | 5
Ejection fraction decreased (Investigations) | 1 | 1
INR increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 7
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 8
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 21
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Nervous system disorders-Other (Nervous system disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 2
Renal calculi (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 7
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 6 | 8
Thromboembolic event (Vascular disorders) | 1 | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=723) | Everolimus (N=740)
Anemia (Blood and lymphatic system disorders) | 151 | 364
Abdominal pain (Gastrointestinal disorders) | 111 | 137
Constipation (Gastrointestinal disorders) | 86 | 86
Diarrhea (Gastrointestinal disorders) | 145 | 289
Dry mouth (Gastrointestinal disorders) | 37 | 55
Dyspepsia (Gastrointestinal disorders) | 46 | 29
Mucositis oral (Gastrointestinal disorders) | 143 | 474
Nausea (Gastrointestinal disorders) | 149 | 208
Vomiting (Gastrointestinal disorders) | 50 | 90
Chills (General disorders) | 25 | 55
Edema limbs (General disorders) | 77 | 170
Fatigue (General disorders) | 366 | 449
Fever (General disorders) | 20 | 61
Pain (General disorders) | 84 | 87
Skin infection (Infections and infestations) | 21 | 45
Upper respiratory infection (Infections and infestations) | 44 | 47
Alanine aminotransferase increased (Investigations) | 69 | 143
Alkaline phosphatase increased (Investigations) | 56 | 104
Aspartate aminotransferase increased (Investigations) | 65 | 159
Blood bilirubin increased (Investigations) | 40 | 12
Cholesterol high (Investigations) | 180 | 396
Creatinine increased (Investigations) | 280 | 323
Lymphocyte count decreased (Investigations) | 27 | 93
Neutrophil count decreased (Investigations) | 21 | 65
Platelet count decreased (Investigations) | 41 | 139
Weight gain (Investigations) | 82 | 33
Weight loss (Investigations) | 17 | 82
White blood cell decreased (Investigations) | 41 | 125
Anorexia (Metabolism and nutrition disorders) | 48 | 134
Hyperglycemia (Metabolism and nutrition disorders) | 268 | 319
Hyperkalemia (Metabolism and nutrition disorders) | 68 | 43
Hypertriglyceridemia (Metabolism and nutrition disorders) | 295 | 419
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 | 59
Hypocalcemia (Metabolism and nutrition disorders) | 27 | 75
Hypokalemia (Metabolism and nutrition disorders) | 16 | 49
Hyponatremia (Metabolism and nutrition disorders) | 52 | 62
Arthralgia (Musculoskeletal and connective tissue disorders) | 118 | 97
Back pain (Musculoskeletal and connective tissue disorders) | 124 | 97
Flank pain (Musculoskeletal and connective tissue disorders) | 55 | 39
Myalgia (Musculoskeletal and connective tissue disorders) | 55 | 74
Pain in extremity (Musculoskeletal and connective tissue disorders) | 90 | 86
Dizziness (Nervous system disorders) | 104 | 112
Dysgeusia (Nervous system disorders) | 48 | 159
Headache (Nervous system disorders) | 156 | 214
Peripheral sensory neuropathy (Nervous system disorders) | 53 | 41
Anxiety (Psychiatric disorders) | 60 | 40
Depression (Psychiatric disorders) | 42 | 32
Insomnia (Psychiatric disorders) | 84 | 86
Urinary frequency (Renal and urinary disorders) | 37 | 46
Cough (Respiratory, thoracic and mediastinal disorders) | 162 | 204
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 80 | 156
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 126
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 45 | 73
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 97
Sore throat (Respiratory, thoracic and mediastinal disorders) | 22 | 70
Dry skin (Skin and subcutaneous tissue disorders) | 77 | 144
Erythema multiforme (Skin and subcutaneous tissue disorders) | 12 | 37
Pruritus (Skin and subcutaneous tissue disorders) | 80 | 147
Rash acneiform (Skin and subcutaneous tissue disorders) | 50 | 218
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 70 | 243
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 53 | 80
Hypertension (Vascular disorders) | 195 | 197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT01120249/Prot_SAP_ICF_000.pdf